CLINICAL TRIAL: NCT00042211
Title: Preventing Depression in Macular Degeneration
Brief Title: Preventing Depression in Patients With Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH061331 (NIH); R01MH061331 (NIH); DATR A4-GPS
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2008-02

CONDITIONS: Depression; Macular Degeneration
Keywords: Depressive Disorder; Blindness; Aged
MeSH Terms: conditions — Depression; Macular Degeneration; Depressive Disorder; Blindness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Problem Solving Treatment
  Interventions: Behavioral: Problem Solving Treatment
- 2 (Active Comparator): Control
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Problem Solving Treatment — Brief Cognitive Behavioral Therapy
  Arms: 1
Behavioral: Control — No treatment control
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a Problem Solving Treatment in preventing depression in elderly patients with age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
AMD is the most common cause of blindness in older adults. The disease limits the ability to read, see familiar faces, and walk independently. Almost 2 million persons (about 5 percent of the U.S. population over age 65) are now affected, and this number will triple by the year 2020. This study will target patients with neovascular AMD (NV-AMD), a form of AMD which can lead to sudden vision loss, substantial disability, and depression. Because depression is itself disabling and not likely to be recognized nor treated by ophthalmologists, preventing depression in people with NV-AMD is important.

Patients are randomly assigned to either PST or a usual care control condition. The primary outcome measure is a DSM-IV diagnosis of depression. Patients are evaluated at baseline, Month 2 (immediately post-intervention), Month 6 (for the primary efficacy analysis), and Month 12 (to evaluate sustained effects). The study will also assess the impact of PST on levels of disability and vision-related quality of life.

ELIGIBILITY:
Inclusion criteria:

* Bilateral macular degeneration
* Visual acuity of 20/40 or worse in better eye
* Residence within 40 miles of Wills Eye Hospital in Philadelphia, PA

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 206 (Actual)
Dates: Start 2001-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Depression | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: barry rovner, md, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Rovner BW, Casten RJ. Activity loss and depression in age-related macular degeneration. Am J Geriatr Psychiatry. 2002 May-Jun;10(3):305-10. PMID 11994218
- [Background] Rovner BW, Casten RJ. Neuroticism predicts depression and disability in age-related macular degeneration. J Am Geriatr Soc. 2001 Aug;49(8):1097-100. doi: 10.1046/j.1532-5415.2001.49215.x. PMID 11555073
- [Background] Rovner BW, Ganguli M. Depression and disability associated with impaired vision: the MoVies Project. J Am Geriatr Soc. 1998 May;46(5):617-9. doi: 10.1111/j.1532-5415.1998.tb01080.x. PMID 9588377
- [Background] Rovner BW, Casten RJ, Tasman WS. Effect of depression on vision function in age-related macular degeneration. Arch Ophthalmol. 2002 Aug;120(8):1041-4. doi: 10.1001/archopht.120.8.1041. PMID 12149057
- [Background] Tasman W, Rovner B. Age-related macular degeneration: treating the whole patient. Arch Ophthalmol. 2004 Apr;122(4):648-9. doi: 10.1001/archopht.122.4.648. No abstract available. PMID 15078685
- [Background] Casten RJ, Rovner BW, Tasman W. Age-related macular degeneration and depression: a review of recent research. Curr Opin Ophthalmol. 2004 Jun;15(3):181-3. doi: 10.1097/01.icu.0000120710.35941.3f. PMID 15118503
- [Background] Casten, R. J., & Rovner, B. W. The role of psychological characteristics in the use and perceived importance of low vision aids. Submitted to the Journal of Vision Impairment and Blindness
- [Background] Rovner BW, Casten R. Stability of visual acuity measurement in depression. Am J Geriatr Psychiatry. 2005 Mar;13(3):255-8. doi: 10.1176/appi.ajgp.13.3.255. PMID 15728758
- [Derived] Rovner BW, Casten RJ, Hegel MT, Leiby BE, Tasman WS. Preventing depression in age-related macular degeneration. Arch Gen Psychiatry. 2007 Aug;64(8):886-92. doi: 10.1001/archpsyc.64.8.886. PMID 17679633